CLINICAL TRIAL: NCT02840903
Title: A Study of the Image Quality in Coronary or Craniocervical CT Angiography With Different Iodine Delivery Rates Using Low Tube Voltage (80 or 100 kV) Imaging in MDCT
Brief Title: A Non-interventional Study to Observe the Computed Tomographic Angiography Image Quality With Different Contrast Media Injection Protocols Under Different Computed Tomography Machines Parameters Setting
Acronym: RIGHT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17811
Record Dates: First submitted 2016-07-06; First posted 2016-07-21 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Angiography; Multidetector Computed Tomography
Keywords: CTA; Computed Tomographic Angiography
MeSH Terms: interventions — iopromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Setting 1 of Iopromide: Craniocervical CTA under below setting: injection rate of iopromide: 4 ml/s, concentration of iopromide = 300 mgI/ml, injection dose of iopromide: 0.8 ml/kg BW, tube voltage = 80 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 2 of Iopromide: Craniocervical CTA under below setting: injection rate of iopromide: 3.2 ml/s, concentration of iopromide = 370 mgI/ml, injection dose of iopromide: 0.65 ml/kg BW, tube voltage = 80 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 3 of Iopromide: Craniocervical CTA under below setting: injection rate of iopromide: 3.2 ml/s, concentration of iopromide = 300 mgI/ml, injection dose of iopromide: 0.8 ml/kg BW, tube voltage = 80 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 4 of Iopromide: Craniocervical CTA under below setting: injection rate of iopromide: 4 ml/s, concentration of iopromide = 370 mgI/ml, injection dose of iopromide: 0.8 ml/kg BW, tube voltage = 100 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 5 of Iopromide: Coronary CTA under below setting: injection rate of iopromide: 4 ml/s, concentration of iopromide = 300 mgI/ml, injection dose of iopromide: 0.8 ml/kg BW, tube voltage = 80 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 6 of Iopromide: Coronary CTA under below setting: injection rate of iopromide: 3.2 ml/s, concentration of iopromide = 370 mgI/ml, injection dose of iopromide: 0.65 ml/kg BW, tube voltage = 80 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 7 of Iopromide: Coronary CTA under below setting: injection rate of iopromide: 3.2 ml/s, concentration of iopromide = 300 mgI/ml, injection dose of iopromide: 0.8 ml/kg BW, tube voltage = 80 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Setting 8 of Iopromide: Coronary CTA under below setting: injection rate of iopromide: 4 ml/s, concentration of iopromide = 370 mgI/ml, injection dose of iopromide: 0.8 ml/kg BW, tube voltage = 100 kvp
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)

INTERVENTIONS:
Drug: Iopromide (Ultravist, BAY86-4877) — 8 settings for CT Angiography as described in group description.

SUMMARY:
The objective of this study is to evaluate the image quality for different iodine delivery rates at different low voltage scanning protocols (80 or 100 kV ) under the modern advanced Multi-Detector Computed Tomography (MDCT) considering the body weight of patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the image quality of different acquisition protocols in patients weighing less than 90 kg using low voltage 80 or 100 kV with a lower Iodine Delivery Rate based on the body weight of the patient, who will undertake coronary or craniocervical CTA (Computed Tomography Angiography) in routine procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom the decision to initiate CTA will be made as per investigator's routine practice.
* Adult patients (age ≥18 years) with a weight ≤ 90 kg.
* Written Informed Consent.

Exclusion Criteria:

* A history of hypersensitivity to iodinated contrast agents.
* Known or suspected hyperthyroidism or pheochromocytoma.
* Atrial fibrillation or any other cardiac arrhythmia that would preclude reliable ECG gating; have severe congestive heart failure (New York Heart Classification IV).
* Pregnant or lactating women.
* Patients participating in another clinical study.
* Patients who underwent PCI (percutaneous coronary intervention) or CABG (coronary artery bypass grafting) before the index CTA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for CT Angiography for examination of the cerebral arteries (suspicion of cerebral artery stenosis or embolism, or suspected carotid pathology) or for examination of the coronary arteries receiving Ultravist at 80 or 100 kV can be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Contrast opacification of the target vascular segments, measured in Hounsfield Units (HU) | Up to 1 week
  Defined as the CT value which can be measured on the CTA images.

SECONDARY OUTCOMES:
Value of CNR (contrast-noise ratio) of the vascular segments | Up to 1 week
  Calculated by the formula: CNR = [Averaged vascular segmental CT value - brain parenchyma (for carniocervical CTA) / perivascular tissues (for Coronary CTA (CCTA)) CT value] / image noise
Value of SNR (signal-noise ratio) of the vascular segments | Up to 1 week
  Calculated by the formula: SNR = Averaged vascular segmental CT value / image noise
Score of visual assessment of the CTA image quality | Up to 1 week
  Subjective visual assessment using a 4-point scale:
  1. Non-diagnostic
  2. Adequate
  3. Good
  4. Excellent
Score of diagnostic confidence of the CTA images | Up to 1 week
  Subjective assessment of diagnostic confidence in the delineation of pathologic findings using a 4-point scale:
  1. Insufficient
  2. Adequate
  3. Good
  4. Excellent
Injected dosage (ml) of the contrast media (CM) | Up to 24 hours
  Can be read from the screen of the CT injector.
Injection rate (ml/s) of the contrast media | Up to 24 hours
  Can be read from the screen of the CT injector.
Value of the Idoine delivery rate (IDR) (unit: mg I/s) | Up to 1 week
  Calculated by the formula:
  IDR (mg I/s) = CM concentration (mg I/ml) * CM injection rate (ml/s)
Value of the volume CT dose index (CTDIvol) (unit: mGy) | Up to 1 week
  A parameter of the radiation dose which can be automatically generated and recorded by the CT machine.
Value of the dose length product (DLP) (unit: mGy*cm) | Up to 1 week
  A parameter of the radiation dose which can be automatically generated and recorded by the CT machine.
Value of the effective dose (organ dose) (unit: mSv) | Up to 1 week
  The effective radiation dose which can be estimated by DLP multiplied by a specific conversion coefficient.
Heart rate of the patients who underwent CCTA before and after the CM injection | Up to 24 hours
  It can be read from the screen of the ECG monitor of the CT machine
Presence of injection pain or discomfort of the patients (Yes/No) | Up to 24 hours
  Assessed by investigators by asking patients if they have injection pain or discomfort.
Number of patients with adverse events / adverse drug reactions | Up to 1 hour
Severity of injection pain or discomfort of the patients | Up to 24 hours
  Assessed by investigators by asking the patients of the severity (mild, moderate, severe) if present.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, China

REFERENCES:
- [Derived] Wang Y, Chen Y, Liu P, Lv W, Wu J, Wei M, Shi D, Wu X, Liu W, Tao X, Hu H, Ma X, Yang X, Xue H, Jin Z. Clinical effectiveness of contrast medium injection protocols for 80-kV coronary and craniocervical CT angiography-a prospective multicenter observational study. Eur Radiol. 2022 Jun;32(6):3808-3818. doi: 10.1007/s00330-021-08505-5. Epub 2022 Feb 1. PMID 35103828